CLINICAL TRIAL: NCT06154980
Title: Randomized Controlled Comparison of Preoperative Ultrasound Guided TLIP Block Versus Intraoperative Non-ultrasound Guided TLIP Block
Brief Title: Randomized Controlled Comparison of Pre-op TLIP vs Intra-op TLIP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Physician is leaving the institution and it will not be continued.
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Daniel K Park, MD, Orthopedic Surgeon, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-189
Record Dates: First submitted 2023-11-16; First posted 2023-12-04 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Pain; Spine Fusion
Keywords: thoracolumbar interfacial plane block; lumbar spine fusion; posterior laminectomy with fusion
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Preoperative Ultrasound TLIP Group (Active Comparator): Participant will receive TLIP in preop with 20cc of 0.2% ropivacaine administered bilaterally, 40cc total. Blocks will be performed under ultrasound guidance with an in-plane technique by a single study investigator.
  Interventions: Procedure: Preoperative Ultrasound TLIP
- Intraoperative TLIP Group (Active Comparator): Participants will receive TLIP with 20cc of 0.2% ropivacaine bilaterally, 40cc total. Blocks will be performed intraoperatively under direct surgical visualization.
  Interventions: Procedure: Intraoperative TLIP

INTERVENTIONS:
Procedure: Preoperative Ultrasound TLIP — TLIP will be performed in preop with 20cc of 0.2% ropivacaine administered bilaterally, 40cc total. Blocks will be performed under ultrasound guidance with an in-plane technique.
  Arms: Preoperative Ultrasound TLIP Group
Procedure: Intraoperative TLIP — TLIP will be performed intraoperatively with 20cc of 0.2% ropivacaine bilaterally, 40cc total. Blocks under direct surgical visualization.
  Arms: Intraoperative TLIP Group

SUMMARY:
Single-center, randomized study will enroll 50 subjects who are scheduled for 1-3 level posterior laminectomy & fusion. Study participants who are eligible for the posterior lumbar laminectomy and fusion procedure will be scheduled and also consented as a part of the study. Participants will be stratified based on age and gender to ensure equal distribution.

DETAILED DESCRIPTION:
This is a single-center, randomized study. The study will enroll 50 subjects who are scheduled for 1-3 level posterior laminectomy & fusion. Potential participants who are eligible for the posterior lumbar laminectomy and fusion procedure will be scheduled as a study participant, consented as a part of the study, and stratified based on age and gender to ensure equal distribution.

For each participant, demographics including age, sex, smoking and alcohol use history, body mass index (BMI), Cranial Cervical Instability (CCI), American Society of Anesthesiology classification (ASA), prior opioid use for pain management, pain levels, function, and prior history of other spinal surgery will be collected prior to surgery. Participants will be randomly assigned to one of two treatment groups: Pre-op ultrasound Thoracolumbar Interfacial Plane Block (TLIP) group or Intra-operative Thoracolumbar Interfacial Plane Block (TLIP) group.

The participant will then undergo the planned 1 to 3 level posterior lumbar laminectomy and fusion procedure.

Post-operative opioid analgesia will be assessed using the Visual Analog Scale (VAS) upon arrival to the post-anesthesia unit (PACU) until discharge and in the outpatient setting. Pain, satisfaction, and opioid analgesia consumption will also be assessed at 2-3 weeks post-operatively, 4-6 weeks post-operatively, and 3 months post-operatively. Pain will be assessed using VAS. Satisfaction will be assessed using a Likert scale. Opioid analgesia is defined as oxycodone, oxymorphone, hydrocodone, hydromorphone, fentanyl, morphine, codeine, methadone, tramadol, and buprenorphine. Opioid consumption will be measured in morphine milligram equivalents (MME).

ELIGIBILITY:
Inclusion Criteria:

* greater than or equal to 18 years of age on the date of service
* require a 1 to 3 level posterior laminectomy with fusion
* compliant with study requirements and outpatient follow-up
* a daily MME less than 25 MME per day in the per-operative period

Exclusion Criteria:

* younger than 18 years of age on the date of service
* does not consent to participating in the program or to be refusal to follow-up at 2-3 weeks, 4-6 weeks, and 3 months post-operatively
* requiring revision surgery at the same level for posterior laminectomy with fusion
* a daily MME score >25 MME/day in the pre-operative period will be excluded
* a positive drug screen for cocaine and/or tetrahydrocannabinol (THC), defined in the standard Corewell Drugs of Abuse Screening as cocaine > 300 ng/mL and cannabinoid > 50 ng/mL-any
* ongoing lawsuits, workers compensation, and litigation will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10-28 (Actual); Primary Completion 2025-10-21 (Actual); Study Completion 2025-10-21 (Actual)

PRIMARY OUTCOMES:
Pain scores at admission to PACU | Baseline (up to 30 days prior to surgery) to PACU admission (immediately post-operative)
  Post operative pain scores will be measured using visual analog scale (VAS) scores at admission to PACU after surgery. The scale is 0-10 with a lower score indicating less pain. A score of 0 indicates no pain and a score of 10 indicates severe pain.
Pain scores at admission to inpatient unit | At inpatient unit admission (within 24 hours after surgery)
  Post operative pain scores will be measured using visual analog scale (VAS) scores at admission to inpatient unit after surgery. The scale is 0-10 with a lower score indicating less pain. A score of 0 indicates no pain and a score of 10 indicates severe pain.
Pain score at discharge from hospital | At hospital discharge (within 3 days of hospital discharge)
  Post operative pain scores will be measured using visual analog scale (VAS) scores at every 8 hours after admission to an inpatient unit until discharge. The scale is 0-10 with a lower score indicating less pain. A score of 0 indicates no pain and a score of 10 indicates severe pain.
Pain score at 2-3 weeks (VAS) | 2-3 weeks after surgery
  Post operative pain scores will be measured using visual analog scale (VAS) scores at the 2-3 week follow-up. The scale is 0-10 with a lower score indicating less pain. A score of 0 indicates no pain and a score of 10 indicates severe pain.
Pain score at 4-6 weeks (VAS) | 4-6 weeks after surgery
  Post operative pain scores will be measured using visual analog scale (VAS) scores at the 4-6 week follow-up. The scale is 0-10 with a lower score indicating less pain. A score of 0 indicates no pain and a score of 10 indicates severe pain.
Pain score at 3 months (VAS) | 3 months after surgery
  Post operative pain scores will be measured using visual analog scale (VAS) scores at the 3 month follow-up. The scale is 0-10 with a lower score indicating less pain. A score of 0 indicates no pain and a score of 10 indicates severe pain.
Pain score at 2-3 weeks (Likert) | 2-3 weeks after surgery
  Post-operative pain will be measured using a 10 point Likert pain score. The scale is 1 - 10 and a lower number indicates less pain. 1 is no pain and 10 is intense pain.
Pain score at 4-6 weeks (Likert) | 4-6 weeks after surgery
  Post-operative pain will be measured using a 10 point Likert pain score. The scale is 1 - 10 and a lower number indicates less pain. 1 is no pain and 10 is intense pain.
Pain score at 3 months (Likert) | 3 months after surgery
  Post-operative pain will be measured using a 10 point Likert pain score. The scale is 1 - 10 and a lower number indicates less pain. 1 is no pain and 10 is intense pain.
Change in pain 24 hours after surgery | 24 hours after surgery
  The change of VAS score from the score at the time of post anesthesia care unit (PACU) arrival to 24 hours after surgery. Pain scores will be measured using visual analog scale (VAS) scores. The scale is 0-10 with a lower score indicating less pain. A score of 0 indicates no pain and a score of 10 indicates severe pain.
Change in back pain at 2-3 weeks | 2-3 weeks after surgery
  The change of VAS score from the score at the time of post anesthesia care unit (PACU) arrival to 2-3 weeks after surgery. Pain scores will be measured using visual analog scale (VAS) scores at the 2-3 week follow-up. The scale is 0-10 with a lower score indicating less pain. A score of 0 indicates no pain and a score of 10 indicates severe pain.
Change in back pain at 4-6 weeks | 4-6 weeks after surgery
  The change of VAS score from the score at the time of post anesthesia care unit (PACU) arrival to 4-6 weeks after surgery. Pain scores will be measured using visual analog scale (VAS) scores at the 4-6 week follow-up. The scale is 0-10 with a lower score indicating less pain. A score of 0 indicates no pain and a score of 10 indicates severe pain.
Change in back pain at 3 months | 3 months after surgery
  The change of VAS score from the score at the time of post anesthesia care unit (PACU) arrival to 3 months after surgery. Pain scores will be measured using visual analog scale (VAS) scores at the 3 month follow-up. The scale is 0-10 with a lower score indicating less pain. A score of 0 indicates no pain and a score of 10 indicates severe pain.
Change in right leg pain at 2-3 weeks | 2-3 weeks after surgery
  The change of VAS score from the score at the time of post anesthesia care unit (PACU) arrival to 2-3 weeks after surgery. Pain scores will be measured using visual analog scale (VAS) scores at the 2-3 week follow-up. The scale is 0-10 with a lower score indicating less pain. A score of 0 indicates no pain and a score of 10 indicates severe pain.
Change in right leg pain at 4-6 weeks | 4-6 weeks after surgery
  The change of VAS score from the score at the time of post anesthesia care unit (PACU) arrival to 4-6 weeks after surgery. Pain scores will be measured using visual analog scale (VAS) scores at the 4-6 week follow-up. The scale is 0-10 with a lower score indicating less pain. A score of 0 indicates no pain and a score of 10 indicates severe pain.
Change in right leg pain at 3 months | 3 months after surgery
  The change of VAS score from the score at the time of post anesthesia care unit (PACU) arrival to 3 months after surgery. Pain scores will be measured using visual analog scale (VAS) scores at the 3 month follow-up. The scale is 0-10 with a lower score indicating less pain. A score of 0 indicates no pain and a score of 10 indicates severe pain.
Change in left leg pain at 2-3 weeks | 2-3 weeks after surgery
  The change of VAS score from the score at the time of post anesthesia care unit (PACU) arrival to 2-3 weeks after surgery. Pain scores will be measured using visual analog scale (VAS) scores at the 2-3 week follow-up. The scale is 0-10 with a lower score indicating less pain. A score of 0 indicates no pain and a score of 10 indicates severe pain.
Change in left leg pain at 4-6 weeks | 4-6 weeks after surgery
  The change of VAS score from the score at the time of post anesthesia care unit (PACU) arrival to 4-6 weeks after surgery. Pain scores will be measured using visual analog scale (VAS) scores at the 4-6 week follow-up. The scale is 0-10 with a lower score indicating less pain. A score of 0 indicates no pain and a score of 10 indicates severe pain.
Change in left leg pain at 3 months | 3 months after surgery
  The change of VAS score from the score at the time of post anesthesia care unit (PACU) arrival to 3 months after surgery. Pain scores will be measured using visual analog scale (VAS) scores at the 3 month follow-up. The scale is 0-10 with a lower score indicating less pain. A score of 0 indicates no pain and a score of 10 indicates severe pain.
Opioid Consumption | PACU arrival through 3 months
  Opioid consumption will be measured in morphine milligram equivalents (MME). This is defined as the amount of milligrams of morphine an opioid dose is equal to. Opioid consumption measured in MME will be collected from PACU through 3 month follow up.

SECONDARY OUTCOMES:
Satisfaction at 3 months | 3 months after surgery
  Satisfaction of surgical outcome will be measured using a 10 point Likert scale. The scale is 1 - 10 and a higher number indicates higher satisfaction with the surgical outcome. 1 is very unsatisfied and 10 is very satisfied.
Satisfaction at 4-6 weeks | 4-6 weeks after surgery
  Satisfaction of surgical outcome will be measured using a 10 point Likert scale. The scale is 1 - 10 and a higher number indicates higher satisfaction with the surgical outcome. 1 is very unsatisfied and 10 is very satisfied.
Satisfaction at 2-3 weeks | 2-3 weeks after surgery
  Satisfaction of surgical outcome will be measured using a 10 point Likert scale. The scale is 1 - 10 and a higher number indicates higher satisfaction with the surgical outcome. 1 is very unsatisfied and 10 is very satisfied.
Number of Adverse Events | Surgery to 3 months
  Adverse events will be collected from the time of surgery through 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Park, MD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Study withdrawn, no individual participant data to share.